CLINICAL TRIAL: NCT01404728
Title: Prospective Longitudinal Evaluation of Vaginal Stenosis and Sexual Function in Women With Pelvic Malignancies Treated With and Without Pelvic Radiation Therapy
Brief Title: Longitudinal Evaluation Study of Vaginal Stenosis With and Without Pelvic Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0454.cc
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Malignancies; Stenosis of Vagina
Keywords: Vaginal length; Sexual dysfunction
MeSH Terms: conditions — Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pelvic Malignancies: Women with Vaginal Stenosis

SUMMARY:
This study evaluates the effects of treatment with a vaginal dilator to reduce vaginal stenosis in women receiving pelvic radiation therapy for pelvic malignancies.

DETAILED DESCRIPTION:
Vaginal stenosis can occur as a result of treatment for pelvic malignancies. Women receiving pelvic radiation therapy using a vaginal dilator 5-7 times per week will have less vaginal stenosis than women using a vaginal dilator fewer times or not at all.

ELIGIBILITY:
Inclusion Criteria:

* Pre and post menopausal women undergoing definitive (not palliative) treatments for a pelvic malignancy, including rectal, endometrial, cervical, or anal canal carcinoma.
* Treatments include radiation therapy, chemotherapy, surgery, or a combination of therapies.
* May have early-stage or locally advanced (node positive) disease.
* Male partners of the female subjects are also consented for this study.

Exclusion Criteria:

* Subject may not have evidence of metastatic disease.
* Prior pelvic radiation therapy
* Prior hysterectomy (not for current diagnosis)
* Diagnosis of prior malignancy, except non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women being treated for pelvic malignancies in the primary care clinic.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2013-01-22 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Observation of a change in vaginal length as measured with a vaginal sound (modified vaginal dilator) | Up to 24 Months
  Observation of change in vaginal length will be measured at baseline (which for the patients in the radiation group will be prior to any pelvic radiation therapy and for patients in the surgery group this will be at the first post-operative visit), as well as in follow-up visits at 3, 6, 12, and 24 months for a total of 5 measurements.
Observation of change in sexual function/satisfaction as measured by the Sexual Adjustment Questionnaire (SAQ) | Up to 24 Months
  The baseline SAQ will be administered prior to radiation therapy for the pelvic malignancy group and it will be administered at the post-operative visit for the surgery only group, and the post-treatment SAQ version will be given at the follow-up visits at 3, 6, 12, and 24 months for a total of 5 measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Fisher, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No